CLINICAL TRIAL: NCT05828264
Title: The Effect of "Quantum-Touch" on Venipuncture Pain, Fear, and Anxiety in Children Aged 7-12 Years Old; Randomized Controlled Study
Brief Title: The Effect of "Quantum-Touch" on Pain, Fear, and Anxiety of the Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Assistant Professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KU
Record Dates: First submitted 2023-04-11; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pain, Acute; Child Behavior; Anxiety and Fear; Venipuncture Site Reaction; Quantum
MeSH Terms: conditions — Acute Pain; Child Behavior; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: this study is an experimental, parallel-group (intervention-control), randomized controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): children in the control group will be received standard care. Control group children will not receive any distraction techniques.
- Quantum Touch (Experimental): The children in the quantum touch groups will received quantum touch application during the venipuncture procedure by the expert nurse
  Interventions: Behavioral: Quantum touch

INTERVENTIONS:
Behavioral: Quantum touch — this group by the nurse who is included in the study and who has a practice certificate before vascular access is established. In this process, the treatment process of the patient will continue and will not create an obstacle. While the child is in a comfortable position (lying or sitting position) during the application, the child's back/shoulder/head will be touched by the practitioner and guantum touch energy will be applied. Then, vascular access will be performed by the nurse included in the study. The child will be asked to rate the level of pain during the procedure with 'FPS-R', the level of fear with 'CDS', and the level of anxiety with 'ÇAS-D'.
  Arms: Quantum Touch

SUMMARY:
This research is a randomized controlled experimental study designed to determine the effect of the Quantum-Touch method applied during the vascular access procedure in children aged 7-12 years, on the level of pain, fear and anxiety in children.

DETAILED DESCRIPTION:
Quantum-Touch was first described by Richard Gordon and Bob Rasmusson in 1978; it activates life force energy by combining various hand positions, various breathing techniques and body awareness exercises. It is applied by directing the formed high energy field to an area of pain, stress or illness through therapeutic touch. Tully found that Quantum Touch in reducing acute and chronic pain; Walton reported that Quantum-Touch application is effective in chronic musculoskeletal pain. It is important to conduct studies with a high level of evidence investigating the effect of Quantum Touch, which is a non-pharmacological method, on pain, fear and anxiety for children of different age groups, which is easily applied during invasive procedures. Based on this information, in this study, which was planned in a randomized controlled and experimental design, it was aimed to determine the effect of the Quantum-Touch method applied during the vascular access procedure in children between the ages of 7-12 on the level of pain, fear and anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* The child and family agree to participate in the research,
* The child's being literate,
* The child is between the ages of 7-12
* The child does not have a chronic and mental health problem.
* No history of sedative, analgesic or narcotic substance use within 24 hours before admission
* Not having a febrile illness at the time of application
* Previous vascular access

Exclusion Criteria:

* The child and family do not agree to participate in the research,
* The child's illiteracy,
* Having a visual and auditory problem,
* The child is less than 7 years old or older than 12 years old
* The child has a chronic and mental health problem
* Failure to open vascular access in a single attempt
* Having a phobia of pain

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale-Revize (FPS-R | One minute after the venipuncture procedure
  This scale consists of 6 facial expressions graded from 0 to 10 according to the presence and severity of pain, and its use is common in children aged 4-16. FPS-R is a valid and reliable individual expression sensitive scale in painful situations in children.
Child Fear Scale | One minute after the venipuncture procedure
  In this scale, the child is shown a picture containing five facial expressions evaluated between 0 and 4. 0 indicates no fear or anxiety; 4 indicates the highest fear and anxiety. These; "0" neutral expression (no anxiety) "1" little fear (very little anxiety) "2" some fear (some anxiety) "3" more fear (more anxiety) "4" highest possible fear (severe anxiety) .
Child Anxiety Scale-State | One minute after the venipuncture procedure
  ÇAS-D is similar to a thermometer with a light bulb at the bottom and horizontal lines at intervals that go up. The scale is aimed at children aged 4-10 years. To measure state anxiety (CAS-D), the child is asked to mark what he feels "right now".

CONTACTS AND LOCATIONS:
Locations (1):
- Remziye Semerci, Edirne, Center, Turkey (Türkiye)